CLINICAL TRIAL: NCT02695368
Title: The Effect of Air-filtration Through a Plasma Chamber on the Incidence of Surgical Site Infections in Orthopaedic Surgery: a Double-blind, Randomized, Controlled Trial
Brief Title: The Effect of Plasma-air-filtration on the Incidence of Surgical Site Infections in Orthopaedic Surgery
Acronym: EPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Max Gordon, M.D., PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EPOS
Record Dates: First submitted 2016-02-09; First posted 2016-03-01 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Orthopaedic Surgery (30 Minutes or Longer)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exposed patients: Plasma-filter on (Experimental): Those operated with Novaerus NV800 on for at least 2 Days prior to index surgery. This Group will also in the analysis be sub-grouped according to measurements prior to study start into:
  * regular operating theater
  * ultra-Clean operating theaters
  Interventions: Device: Novaerus NV800 on
- Unexposed patients: Plasma-filter off (Experimental): Those with Novaerus NV800 off for at least 2 Days prior to index surgery
  Interventions: Device: Novaerus NV800 off
- Mixed patients: Plasma-filter on or off (Experimental): Those receiving multiple surgeries in different theaters with Novaerus NV800 on or off status will belong to a mixed Group.
  Interventions: Device: Novaerus NV800 on or off

INTERVENTIONS:
Device: Novaerus NV800 on — The air-cleaner sterilizes the air particles through a plasma chamber. Air in the operating theatre is pumped through the chamber (80 - 380 m3/Hr) and by using a small current it transforms the gas in the vicinity of the electrode into plasma and eradicates any bacteria that pass through. The air-cleaner has to have been turned on for at least 2 days prior to the surgical intervention.
  Arms: Exposed patients: Plasma-filter on
Device: Novaerus NV800 off — The machine decribed above is running but the plasma filter chamber isn't active, i.e. the placebo group.
  Arms: Unexposed patients: Plasma-filter off
Device: Novaerus NV800 on or off — Patients with multiple surgeries that have been operated during both periods when the apparatus has been on and off will belong to this mixed group.
  Arms: Mixed patients: Plasma-filter on or off

SUMMARY:
The study is a multicenter, double-blind, randomized, controlled trial conducted at six major university and teaching hospitals with a catchment population of approximately 2 million. In the current study it has been hypothesized that a non-invasive air cleaner utilizing a plasma chamber can significantly reduce the incidence of surgical site infections (SSIs).

DETAILED DESCRIPTION:
Despite operating in clean theaters, surface sterilization, and antibiotics, surgical site infections (SSI) after orthopaedic surgery have an estimated incidence of 1-4%. This feared complication is associated with long-term antibiotics, repeated surgeries, prolonged hospital stays, economic burden and a poorer end result for individual patients. It is therefore of great importance to prevent SSI.While skin bacteria and contaminated surfaces have generally been claimed to be the main cause of infections, there are estimates that approximately 20% of hospital-acquired infections are air-transmitted, making this an interesting intervention target. Novaerus is an air-cleaner that sterilizes the air particles through a plasma chamber. Air in the operating theatre is pumped through the chamber (80-380 m3/Hr) and by using a small current it transforms the gas in the vicinity of the electrode into plasmaand eradicates any bacteria that pass through.The small size of the machine allows it to fit into any operating theater without interfering with existing equipment. This technology can reduce the number of colony forming units (CFU) when in hospital settings. In non-randomized settings it has been correlated to reduced respiratory infections, reduced personnel sick-leave, and absence of severe infectious outbreaks. Its effect has not been validated in randomized controlled trials. Both local and national registry data will be used according to availability.

ELIGIBILITY:
Inclusion Criteria:

* All patients that undergo a 30 minute or longer orthopaedic surgery

Exclusion Criteria:

* The following surgeries will be excluded: already infected surgical site, defined as: ICD-codes indicating infection, Open fractures, Traumatic wounds, Vacuum assisted wound therapy
* Patients that have had antibiotics prescribed 2 weeks or less prior to surgery
* Patients that have actively marked their hospital charts with an added privacy notice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45000 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with surgical site infection after orthopaedic surgery, defined as any of the following: using antibiotics targeting Staphylococcus aureus, having ICD-codes or surgery codes indicating postoperative infection. | Within 12 weeks after surgery
  All definitions are merged into one binary outcome measure as "any(No. > 0)"

SECONDARY OUTCOMES:
Patients using any antibiotics after surgery | Two treatment days or more during the first 30 postoperative days
  This is identified either via hospital information system or from the national drug registry. Usage is defined as withdrawal or prescription of a drug with ATC code within the J01 group.
Number of days with antibiotics | During the first 30 postoperative days
  This is identified either via hospital information system or from the national drug registry. Usage is defined as withdrawal or prescription of a drug with ATC code within the J01 group. Number of days is deduced from the prescribed dosage or if not present the average daily dosage for that particular drug is used.
Patients using any antibiotics after surgery | Two treatment days or more during the first 90 postoperative days
  This is identified either via hospital information system or from the national drug registry. Usage is defined as withdrawal or prescription of a drug with ATC code within the J01 group.
Number of days with antibiotics | Two treatment days or more during the first 90 postoperative days
  This is identified either via hospital information system or from the national drug registry. Usage is defined as withdrawal or prescription of a drug with ATC code within the J01 group. Number of days is deduced from the prescribed dosage or if not present the average daily dosage for that particular drug is used.
Death | during the first 2 postoperative years
  Any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Max Gordon, M.D, PhD, Principal Investigator — Danderyd Hospital, Stockholm, Sweden
Locations (1):
- Danderyds Sjukhus AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persson A, Atroshi I, Tyszkiewicz T, Hailer NP, Lazarinis S, Eisler T, Brismar H, Mukka S, Kernell PJ, Mohaddes M, Skoldenberg O, Gordon M. Effect of Plasma Air Purifiers on Infection Rates in Orthopedic Surgery. NEJM Evid. 2025 Apr;4(4):EVIDoa2400289. doi: 10.1056/EVIDoa2400289. Epub 2025 Mar 25. PMID 40130977
- [Derived] Persson A, Atroshi I, Tyszkiewicz T, Hailer N, Lazarinis S, Eisler T, Brismar H, Mukka S, Kernell PJ, Mohaddes M, Skoldenberg O, Gordon M. EPOS trial: the effect of air filtration through a plasma chamber on the incidence of surgical site infection in orthopaedic surgery: a study protocol of a randomised, double-blind, placebo-controlled trial. BMJ Open. 2022 Feb 3;12(2):e047500. doi: 10.1136/bmjopen-2020-047500. PMID 35115346